CLINICAL TRIAL: NCT00317135
Title: Assess Reactogenicity and Safety of GSK Biologicals' Tritanrix™-HepB/Hib-MenAC Compared to Tritanrix™-HepB/Hiberix™ (Control) in Healthy Infants (2,4,6 Months Age), After a Hepatitis B Birth Dose
Brief Title: Safety Study of a Vaccine Against Meningitis in Infants ( 2,4 & 6 Months Age) After a Birth Dose of Hepatitis B.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 759346/004
Record Dates: First submitted 2006-02-15; First posted 2006-04-24 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Diphtheria; Hepatitis B; Whole Cell Pertussis; Haemophilus Influenzae Type b; Tetanus
MeSH Terms: conditions — Diphtheria; Hepatitis B; Haemophilus Infections; Tetanus

ARMS (4):
- Hib-MenAC Lot 1 Group (Experimental): Healthy male or female subjects aged 56 to 83 days of age at the time of the first study vaccine dose, with previous hepatitis B vaccine at birth, received Tritanrix-HepB combined vaccine mixed extemporaneously with Meningitec conjugate vaccine Lot 1 at 2, 4 and 6 months of age as an intramuscular injections in the anterolateral part of the left thigh.
  Interventions: Biological: Tritanrix-HepB/Meningitec conjugate vaccine
- Hib-MenAC Lot 2 Group (Experimental): Healthy male or female subjects aged 56 to 83 days of age at the time of the first study vaccine dose, with previous hepatitis B vaccine at birth, received Tritanrix-HepB combined vaccine mixed extemporaneously with Meningitec conjugate vaccine Lot 2 at 2, 4 and 6 months of age as an intramuscular injections in the anterolateral part of the left thigh.
  Interventions: Biological: Tritanrix-HepB/Meningitec conjugate vaccine
- Hib-MenAC Lot 3 Group (Experimental): Healthy male or female subjects aged 56 to 83 days of age at the time of the first study vaccine dose, with previous hepatitis B vaccine at birth, received Tritanrix-HepB combined vaccine mixed extemporaneously with Meningitec conjugate vaccine Lot 3 at 2, 4 and 6 months of age as an intramuscular injections in the anterolateral part of the left thigh.
  Interventions: Biological: Tritanrix-HepB/Meningitec conjugate vaccine
- Hiberix Group (Active Comparator): Healthy male or female subjects aged 56 to 83 days of age at the time of the first study vaccine dose, with previous hepatitis B vaccine at birth, received Tritanrix-HepB vaccine mixed extemporaneously with conjugate vaccine Hiberix at 2, 4 and 6 months of age as intramuscular injection in the anterolateral part of the thigh.
  Interventions: Biological: Tritanrix/Hiberix vaccine

INTERVENTIONS:
Biological: Tritanrix-HepB/Meningitec conjugate vaccine — The full content of two monodose vials of Tritanrix-HepB vaccine vial was extracted and injected into the vial containing the lyophilized Meningitec (5/5/5) vaccine. The vial was agitated until the lyophilized vaccine pellet had completely dissolved. The reconstituted mixed vaccines were used promptly after reconstitution (within 30 minutes): one dose of 0.5 ml of the reconstituted Tritanrix- HepB/Meningitec vaccine was withdrawn from the vial and administered, the needle was changed before injection
  Other Names: DTPw-HBV/Hib-MenAc conjugate vaccine
  Arms: Hib-MenAC Lot 1 Group; Hib-MenAC Lot 2 Group; Hib-MenAC Lot 3 Group
Biological: Tritanrix/Hiberix vaccine — The full content of the Tritanrix-HepB vaccine vial was extracted and injected into the vial containing the lyophilized Hiberix vaccine. The vial was agitated until the lyophilized vaccine pellet had completely dissolved. The reconstituted mixed vaccines were used promptly after reconstitution (within 30 minutes): the full volume of the mixed vaccines was withdrawn from the vial, the needle was changed before injection.
  Other Names: DTPw-HBV/Hib vaccine
  Arms: Hiberix Group

SUMMARY:
The purpose of this study is to compare the reactogenicity & safety of Tritanrix™-HepB/Hib-MenAC vaccine to the international standard of care, Tritanrix™-HepB/Hiberix™.

DETAILED DESCRIPTION:
Randomized study with four groups to receive one of the following vaccination regimens after a dose of hepatitis B vaccine given at birth:

- One of the 3 lots of GSK Biologicals' Hib-MenAC mixed with GSK Biologicals' Tritanrix™-HepB (3 different groups) - GSK Biologicals' Tritanrix™-HepB/Hiberix™

ELIGIBILITY:
Inclusion criteria at study entry:

* Healthy infants aged less than or equal to 3 days of age, written informed consent obtained from the parents, born after a gestation period of 36 to 42 weeks.

Exclusion criteria at study entry:

* Any confirmed immunodeficient condition, based on medical history & physical examination.
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Acute disease at the time of enrolment.

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2003-12-11; Primary Completion 2004-10-23 (Actual); Study Completion 2004-10-23 (Actual)

PRIMARY OUTCOMES:
Occurrence of fever > 38.5°C(axillary) during the 4-day follow-up period after dose 1 | Days 0-3 post dose 1
Occurrence of fever > 38.5°C(axillary) during the 4-day follow-up period after dose 2 | Days 0-3 post dose 2
Occurrence of fever > 38.5°C(axillary) during the 4-day follow-up period after dose 3 | Days 0-3 post dose 3

SECONDARY OUTCOMES:
Occurrence of solicited symptoms other than fever >38.5°C (axillary) during the 4-day follow-up period after each dose | Days 0-3 after each dose
Occurrence of unsolicited symptoms during the 31-day follow-up period after each dose | Day 0-30 after each dose
Occurrence of serious adverse events during the entire study period | Day 0 up to Month 5

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, City of Muntinlupa, Philippines